CLINICAL TRIAL: NCT05021107
Title: Effects Of Fascial Distortion Model With And Without Neck Isometrics In Patients With Cervical Spine Overload
Brief Title: Fascial Distortion Model With And Without Neck Isometrics In Patients With Cervical Spine Overload
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0119 Adeel
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Fascial Distortion Model with neck isometrics
  Interventions: Other: FDM with isometrics
- Group B (Active Comparator): Fascial Distortion Model with neck isometrics
  Interventions: Other: FDM without isometrics

INTERVENTIONS:
Other: FDM with isometrics — FDM with isometrics will be done
  Arms: Group A
Other: FDM without isometrics — FDM without isometrics will be done
  Arms: Group B

SUMMARY:
Cervical spine pain is the one the most common musculoskeletal disorder and spinal overload is one of the major causes. Forward tilting of every inch of head increases load on the cervical spine and is referred as cervical spine overload. Persistent overloading and overburdening results in radiation of pain, weakness of muscles and limitation in joint range.

Psychological factors are also play role in acute, sub-acute or chronic neck pain. Treatment commonly used for this pain is NSAID, physiotherapy interventions (mobilisation, manipulation, TENS, ultrasound, stretching, isometrics and FDM) and awareness about posture. FDM was established in 1991 by Stephan Typaldos and it recommends that musculoskeletal ailments are due to disruption in fascia. There are 6 diverse proposed facial distortions and diagnosis in this model i.e., trigger band, herniated trigger band, folding distortion, continuum distortion, tectonic fixation and cylinder distortion. Main purpose of this randomised clinical trial will be to find out the effects of fascial distortion model with and without neck isometrics in patients with cervical spine overload.

Patients will be recruited into study by consecutive sampling technique and after that patients will be allocated to the groups by random sampling assignment. NPRS, NDI and goniometer will be used as data measuring tool. Treatment will be given to 2 groups. One group will get treatment of only FDM and other group will get treatment of FDM and neck isometrics as well. Treatment will be given two times a week for 4weeks and duration of the session will be of 30 minutes. After collecting data from defined study setting, data will be entered and analyzed by using Statistical Package for the Social Sciences (SPSS) for Windows software, version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be use within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria:

   * Trigger band pain pattern
   * Age limit 20 to 30 years.
   * Male and female
   * Pain in the cervical spine
   * Limited cervical ROM
   * Uneasiness while working in a sitting posture for 4 hours but no abnormal neurological findings

Exclusion Criteria:

* Progressive degeneration of spine (spondylosis)
* Previous cervical spine injuries
* Congenital and developed spine deformities (scoliosis)

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
NPRS | 4 weeks
  will be used for pain measurement. It is a unitdimensional 11 point scale (0-10) with measure of pain intensity with High test-retest reliability of r = 0.96 and validity correlations range from 0.86 to 0.95.
NDI | 4 weeks
  will be used to check neck disability. Item scores range from 0 to 5, and the total score is a total of the item scores (possible range 0 (no pain) - 100 (maximal pain)
Goniometer | 4 weeks
  to measure range

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Sanabil Health Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sipko T, Biec E, Demczuk-Wlodarczyk E, Ciesielska B. Mobility of cervical spine and postural equilibrium in patients with spinal overload syndrome. Ortop Traumatol Rehabil. 2007 Mar-Apr;9(2):141-8. English, Polish. PMID 17514162
- [Background] Dasgupta S, Rozario JE. Troika of Posture, Occlusion and Airway. Indian J Otolaryngol Head Neck Surg. 2020 Mar;72(1):49-54. doi: 10.1007/s12070-019-01734-7. Epub 2019 Sep 11. PMID 32158655
- [Background] Mysliwiec A, Saulicz E, Kuszewski M, Kokosz M, Wolny T. Assessment of the influence of Saunders traction and transcutaneous electrical nerve stimulation on hand grip force in patients with neck pain. Ortop Traumatol Rehabil. 2011 Jan-Feb;13(1):37-44. doi: 10.5604/15093492.933786. English, Polish. PMID 21393647
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245